CLINICAL TRIAL: NCT03541824
Title: Reducing Suicide Risk Associated With Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Pamela Keel, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10274002
Record Dates: First submitted 2017-12-03; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Eating Behavior; Self Harm; Weight Loss
MeSH Terms: conditions — Feeding Behavior; Self-Injurious Behavior; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Acceptance Program (Experimental): The Body Acceptance Program (BAP) is the active condition. Participants engage in an online intervention during which they complete online and offline activities designed to challenge the appearance-ideal.
  Interventions: Behavioral: Body Acceptance Program
- Waitlist control (No Intervention): Participants in the waitlist control group completed baseline and follow-up assessments with no intervention.

INTERVENTIONS:
Behavioral: Body Acceptance Program — The Body Acceptance Program is a mixed-gender modification of the eBody Project, an online intervention in which cognitive dissonance principals are used to reduce eating pathology.
  Other Names: eBody Project
  Arms: Body Acceptance Program

SUMMARY:
The purpose of this study is to examine the efficacy of an intervention aimed at promoting a healthy lifestyle and reducing risk factors associated with eating pathology, nonsuicidal self-injury, and suicidal behavior. We are also interested in assessing whether this intervention has the potential to prevent future symptoms of eating problems and self-harm urges and behaviors. The broader goal of this research is to identify factors that may help us better understand the prevention of self-harm behaviors and develop more effective treatments for these problems.

DETAILED DESCRIPTION:
The current study was designed as a proof-of-concept study to test the association between weight suppression (WS; difference between one's highest and lowest weight) and non-suicidal self-injury (NSSI). Previous research has found an association between current WS and lifetime NSSI and that this association was mediated by depressive symptoms and drive for thinness. The current study therefore modified an existing online cognitive dissonance-based program (the e-Body Project) using mixed gender content (from the Body Project 4 All scripts) to target posited mediators, i.e., depressive symptoms and weight and shape concerns, in a sample of individuals with WS and engagement in current NSSI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* At least 5 pounds weight suppression
* Engaged in non-suicidal self-injury at least once in past month

Exclusion Criteria:

* Indicated being "sure" of suicide attempt on eligibility screener
* Live outside of the United States
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Self-Injurious Thoughts and Behaviors Interview-Short Form (self-report) at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Self-harm frequency and likelihood

SECONDARY OUTCOMES:
Change from baseline on the "Body Esteem Scale: Appearance" subscale at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Feelings about one's appearance; scores are summed and range from 0-40, higher scores indicate greater appearance esteem
Change from baseline on the "Body Esteem Scale: Weight" subscale at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Feelings about one's weight; scores are summed and range from 0-32, higher scores indicate greater weight esteem
Change from baseline on the "Body Esteem Scale: Attribution" subscale at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Feelings about one's characteristics; scores are summed and range from 0-20, higher scores indicate greater self-esteem
Change from baseline on the Beck Depression Inventory II at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Depressive symptoms
Change from baseline on the Body Shape Questionnaire (8-item version #3) at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Assessment of weight and shape concerns
Change from baseline on the Positive and Negative Affect Schedule at follow-up | Pre-assessment and post-assessment (after intervention or two weeks from baseline)
  Captures current positive and negative affect

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Keel, Ph.D., Principal Investigator — Florida State University

IPD SHARING:
Plan to Share IPD: Yes
Participants' responses to measures collected during the study will be shared with the funding body, the Military Suicide Research Consortium, as part of their Core Data Elements project, a centralized database of data from all MSRC funded projects. All participant responses are deidentified and are uploaded to the MSRC through a secure upload.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and informed consent forms will be shared during and after study recruitment. Participants' responses to measures collected during the study will be shared at the end of participant completion.
Access Criteria: Once data is uploaded to the Core Data Element (CDE) project, it may be combined with data from other projects for greater power to conduct statistical analyses, including, but not limited to, regression analyses and scale development. The following link (https://msrc.fsu.edu/members/request-access-msrc-database) describes steps that investigators must take in order to access the data. In addition, the study protocols and consent forms are reviewed and approved by the Department of Defense Human Research Protection Office (HRPO) throughout the study.

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617